CLINICAL TRIAL: NCT07144176
Title: An Open-label, Randomized, Fasting, Single-dose, Two-treatment, Two-period, Crossover, Phase 1 Clinical Trial to Compare and Evaluate the Pharmacokinetics and Safety of "DWJ1511" and "DWC202501" in Healthy Adult Volunteers
Brief Title: PK and Safety Comparison of DWJ1511 and DWC202501 in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWJ1511101
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A(RT) (Experimental): 30 Subjects, Cross-over, Single dose DWC202501 on period 1, Single dose of DWJ1511 on period 2
  Interventions: Drug: DWJ1511; Drug: DWC202501
- B(TR) (Active Comparator): 30 Subjects, Cross-over, Single dose DWJ1511 on period 1, Single dose of DWC202501 on period 2
  Interventions: Drug: DWJ1511; Drug: DWC202501

INTERVENTIONS:
Drug: DWJ1511 — Test drug: DWJ1511
Drug: DWC202501 — Comparator: DWC202501

SUMMARY:
PK and Safety Comparison of DWJ1511 and DWC202501 in Healthy Volunteers

DETAILED DESCRIPTION:
This is an open-label, randomized, single-dose, two-treatment, two-period, crossover, phase 1 clinical trial conducted under fasting conditions to compare and evaluate the pharmacokinetics (PK) and safety of DWJ1511 and DWC202501. in healthy adult volunteers. Participants will receive both study drugs in separate periods, with a washout interval between administrations. The study aims to assess PK parameters and monitor safety through clinical evaluations and laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged ≥19 years and <65 years at the time of screening
* Body mass index (BMI) between 18 and 30 kg/m² (BMI = weight [kg] / height [m]²)

Exclusion Criteria:

* Subjects who have participated in a bioequivalence study or any other clinical trial and have received an investigational product within 6 months prior to the first administration.
* Subjects who have donated whole blood within 8 weeks prior to the first administration, donated blood components within 2 weeks prior to the first administration, or received a blood transfusion within 4 weeks prior to the first administration.
* Subjects with a history of gastrointestinal surgery that may affect drug absorption (appendectomy and hernia repair are not exclusionary).

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma drug concentration-time curve [AUCt] | 0-12 Hours
  Area under the plasma drug concentration-time curve [AUCt] of DWJ1511 and DWC202501
Maximum plasma concentration [Cmax] | 0-12 Hours
  Maximum plasma concentration [Cmax] of DWJ1511 and DWC202501

SECONDARY OUTCOMES:
Area under the plasma drug concentration-time curve from time 0 to infinity [AUCinf] | 0-12 Hours
  Area under the plasma drug concentration-time curve from time 0 to infinity [AUCinf] of DWJ1511 and DWC202501

CONTACTS AND LOCATIONS:
Locations (1):
- H Plus Yangji Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No